CLINICAL TRIAL: NCT04577703
Title: Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of Ningetinib (CT053PTSA) in Patients With Advanced Solid Tumors: A Phase I, Single-arm, Single-center, Open-label, Dose-escalation Study
Brief Title: First-In-Human Phase I Trial of Ningetinib ( CT053PTSA ) in the Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DCT053-12-003
Record Dates: First submitted 2020-09-16; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT053PTSA (dose escalation) (Experimental): Patients were treated in 5 dose cohorts of 15 mg, 30 mg, 60 mg, 100 mg, and 150 mg QD capsules.
  Patients receive treatment with CT053PTSA once on Cycle 0 Day 1 following a 7-day treatment-free withdrawal period to observe the safety and pharmacokinetic of CT053PTSA.
  After that, Patients receive treatment with CT053PTSA per orally, beginning on Cycle 1 Day 1 for 28 day following a 7-day treatment-free withdrawal period to observe efficacy of CT053PTSA and determine to continue taking medicine or not. Each cycle had 28 days.
  Interventions: Drug: CT053PTSA

INTERVENTIONS:
Drug: CT053PTSA — CT053PTSA will be administered daily in fasting state
  Other Names: Ningetinib

SUMMARY:
This is a phase I, single-arm, single-center, open-label, dose-escalation Study evaluating the safety and efficacy of CT053PTSA in patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a dose-escalation study. The primary purpose is to determine the dose limiting toxicity (DLT), maximum tolerated dose (MTD) and recommend doses and regimen of CT053PTSA for further studies.

ELIGIBILITY:
Inclusion Criteria:

- A. Subjects with advanced solid tumors confirmed by histologically or cytologically that are refractory to current treatment or for which there is not a current standard of care B. Toxicity recovered to NCI CTCAE v.4.0 Grade ≤1 from previous treatments (chemotherapy, radiotherapy or surgery) C. ECOG performance status (PS) 0 or 1 D. Life expectancy of ≥ 12 weeks E. Adequate organ function

1. Hemoglobin > 9 g/dL (SI Units: 90 g/L) without transfusion support or growth factors; Platelet count ≥ 100 × 10^9/L; Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L without growth factor support.
2. AST/SGOT and/or ALT/SGPT≤ 2.5 × upper limit of normal (ULN) or ≤ 5.0× ULN if liver metastases are present; serum bilirubin ≤ 1.5×ULN
3. Serum creatinine ≤ 1.5×ULN
4. Blood potassium≥ 3.0 mmol/L; serum calcium≥2.0 mmol/L
5. Fasting serum triglyceride level≤5.7 mmol/L
6. Asymptomatic abnormal serum amylase≤1.5×ULN
7. Serum lipase≤ ULN
8. INR≤ 1.5×ULN；APTT≤ 1.5×ULN； PT ≤ 1.5×ULN

Exclusion Criteria:

1. Chemotherapy, immunotherapy, radiotherapy, or major surgery within 4 weeks prior to study treatment
2. Nitrosourea, anthracyclinea and mitomycin chemotherapy within 6 weeks prior to study treatment
3. Had received live vaccine within 4 weeks prior to study treatment
4. Had received any investigational agent from other clinical study within 4 weeks prior to study treatment or are currently participating in other clinical trials
5. Previous treatment with any other c-MET inhibitor or HGF inhibitor
6. Symptomatic, untreated or unstable central nervous system metastases
7. Spinal cord compression, carcinomatous meningitis or leptomeningeal diseaseonly (patient are only permitted if treated, asymptomatic and stable for at least 4 weeks prior to start of study treatment)
8. Patients with hypertension that can't be well controlled by drugs (systolic blood pressure> 140 mmHg or diastolic blood pressure> 90 mmHg)
9. Doppler ultrasound evaluation：Left ventricular ejection fraction < 50%
10. Grade ≥ 2 of arrhythmia (assessed by NCI CTCAE 4.0), or symptomatic bradycardia, or male with QTCF > 450 ms or female with QTCF > 470 ms, or patients with a history of torsion or congenital QT prolonged syndrome long QT syndrome
11. Certain factors that would preclude adequate absorption of CT053PTSA (eg. unable to swallow, chronic diarrhea, intestinal obstruction)
12. Significant hemoptysis within 2 months prior to enrollment, or a daily hemoptysis volume is 2.5 ml or above
13. Patients with evidence of bleeding tendency, including the following cases: gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ and above; or melena or hematemesis within 2 months; or visceral bleeding that may occur considered by investigator
14. History of immunodeficiency, or other acquired or congenital immunodeficiency, or history of organ transplantation
15. Any disease of the following bellowed within 12 months prior to administration: Myocardial infarction, severe angina, or unstable angina, coronary or peripheral artery bypass graft, congestive heart failure, or cerebrovascular events (including transient ischemic attack)
16. Pulmonary embolism within 6 months prior to administration
17. Active infection of hepatitis B, hepatitis C, or infection of HIV
18. Undergone a bone marrow or solid organ transplant.
19. Patients with severe retinopathy or exfoliation in the investigator's judgment
20. Patients need to be supplemented with stem cells before receiving large dose chemotherapy (except for myeloma or lymphoma)
21. History of thyroid dysfunction, and the thyroid function cannot be maintained at the normal range with drugs.
22. Anticoagulants, vitamin K antagonists, other anti-tumor drugs and drugs that prolong the QT interval are not allowed.
23. Serious electrolyte imbalance in the investigator's judgment
24. Pregnant or lactating woman
25. Any other reason the investigator considers the patient is not suitable to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02-08 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2015-12-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Cycle 0 Day 1 to Cycle 1 Day 28
  The maximum tolerated dose (MTD) of the CT053PTSA will be determined according to incidence of dose-limiting toxicity (DLT) assessed by NCI CTCAE v4.0

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of CT053PTSA_Cmax | Cycle 0 Day 1 to Cycle 1 Day 28
  To evaluate the Pharmacokinetics (PK) of CT053PTSA with Maximum observed plasma concentration (Cmax)
Pharmacokinetics (PK) of CT053PTSA_Tmax | Cycle 0 Day 1 to Cycle 1 Day 28
  To evaluate the Pharmacokinetics (PK) of CT053PTSA with Time of maximum observed plasma concentration (Tmax).
Pharmacokinetics (PK) of CT053PTSA_AUC | Cycle 0 Day 1 to Cycle 1 Day 28
  To evaluate the Pharmacokinetics (PK) of CT053PTSA with Area under the plasma concentration time curve (AUC).
Efficacy of CT053PTSA_ORR | up to approximately 36 months
  To assess overall response rate (ORR) for patients treated CT053PTSA.
Efficacy of CT053PTSA_DCR | up to approximately 36 months
  To assess disease control rate (DCR) for patients treated CT053PTSA.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No